CLINICAL TRIAL: NCT01113190
Title: Optimizing SBIRT for Drug-Using Patients in an Inner-City Emergency Department
Brief Title: Healthier You: Optimizing Screening, Brief Interventions, and Referral to Treatment (SBIRT) in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frederic C. Blow, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: DA026029; R01DA026029 (NIH)
Record Dates: First submitted 2010-04-20; First posted 2010-04-29 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- CBI in ED with AMET at 3 months (Active Comparator): computer-delivered brief intervention (CBI) at baseline with adapted motivational enhancement therapy-AMET at 3 months
  Interventions: Behavioral: Computer-delivered Brief Intervention (CBI); Behavioral: Adapted Motivational Enhancement Therapy (AMET)
- CBI in ED with EUC at 3 months (Active Comparator): computer-delivered brief intervention (CBI) at baseline with enhanced usual care-EUC at 3 months
  Interventions: Behavioral: Computer-delivered Brief Intervention (CBI); Behavioral: Enhanced Usual Care (EUC)
- IBI in ED with AMET at 3 months (Active Comparator): intervener-delivered brief intervention (IBI) at baseline with adapted motivational enhancement therapy-AMET at 3 months
  Interventions: Behavioral: Intervener-delivered Brief Intervention (IBI); Behavioral: Adapted Motivational Enhancement Therapy (AMET)
- IBI in ED with EUC at 3 months (Active Comparator): intervener-delivered brief intervention (IBI) at baseline with enhanced usual care-EUC at 3 months
  Interventions: Behavioral: Intervener-delivered Brief Intervention (IBI); Behavioral: Enhanced Usual Care (EUC)
- EUC in ED with AMET at 3 months (Active Comparator): enhanced usual care (EUC) at baseline with adapted motivational enhancement therapy-AMET at 3 months
  Interventions: Behavioral: Adapted Motivational Enhancement Therapy (AMET); Behavioral: Enhanced Usual Care (EUC)
- EUC in ED with EUC at 3 months (Active Comparator): enhanced usual care (EUC) at baseline with EUC at 3 months
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Computer-delivered Brief Intervention (CBI) — The multimedia, interactive Computer BI (CBI) condition will be delivered using tablet computers. The content and format will be easily negotiated by participants. The proposed CBI condition will use actors with 'green screen' to deliver scripted therapist content that will be highly tailored to individual responses. 'Green screens' are standard recording formats that allow for inserting engaging background and other overlays onto recorded material. This program will be viewed on a touch screen tablet computer with audio delivered via headphones. The CBI will be designed in a therapist video-delivered interactive style, that provides tailoring options for reviewing patient goals, providing feedback regarding substance use patterns and consequences, completing a "decisional balance" exercise, and formulating a change plan. It requires active participation and is not a passive video that is merely viewed.
  Arms: CBI in ED with AMET at 3 months; CBI in ED with EUC at 3 months
Behavioral: Intervener-delivered Brief Intervention (IBI) — IBI is a 30-minute intervention session with a master's-level clinician. The interventions will include FRAMES (Miller & Rollnick, 2002): personalized Feedback (regarding substance use, risk factors), emphasis on Responsibility for change, Advice, Menu of options, Empathic clinical behaviors, and support of Self-Efficacy regarding making changes. The interventions are designed to address the primary target behavior of drug use, and will include a tailored review of participants' goals/values, feedback regarding their present substance use patterns and consequences, developing a discrepancy between their substance use and ability to meet goals and values through a decisional balance exercise, and formulation of a "change plan" tailored for each participant. IBI will be highly individualized to participants' goals, values and substance use, and will will follow similar session outlines and length of delivery as the CBI sessions.
  Arms: IBI in ED with AMET at 3 months; IBI in ED with EUC at 3 months
Behavioral: Adapted Motivational Enhancement Therapy (AMET) — This session will have a similar general outline to the sessions conducted in the ED, including a review of participants' goals and values, and a review of their substance use and consequences, use of decisional balance exercises as indicated, and review and modification of their change plan. For the AMET intervention, the intervener (at least master's level) will conduct a single session (~30-45 minutes) in the community (HMC ED or our community research office). The therapist will be able to tailor their approach to each individual's needs and motivational state.
  Arms: CBI in ED with AMET at 3 months; EUC in ED with AMET at 3 months; IBI in ED with AMET at 3 months
Behavioral: Enhanced Usual Care (EUC) — The EUC group will receive brief advice to change their drug use, as well as a booklet including information on community support groups, location of substance use treatment centers, mental health services, suicide prevention hotlines, risk of injecting drugs including HIV and hepatitis and HIV prevention and testing information.
  Arms: CBI in ED with EUC at 3 months; EUC in ED with AMET at 3 months; EUC in ED with EUC at 3 months; IBI in ED with EUC at 3 months

SUMMARY:
Screening, brief interventions, and referral to treatment (SBIRT) for drug use/abuse offers opportunities for early detection, brief intervention/treatment, and substance use treatment referrals for patients in medical settings. Although SBIRT components, particularly screening and brief interventions, have been shown to be effective strategies for addressing alcohol misuse in primary care, data are limited on using all of the components of SBIRT for drug-using patients, particularly in the Emergency Department (ED). Further, because of the often chaotic environment of EDs, many logistical and practical impediments exist for the adoption of the entire SBIRT model in this setting.

DETAILED DESCRIPTION:
The proposed study will use computerized screening using touch screen computer tablets with audio (~4,900 patients) and will test intervention strategies in a two-factorial design (3x2). Specifically, 900 patients aged 18-60 in an inner-city ED who screen positive for drug use in the past 3 months will be randomized to the combinations of three ED-based conditions (computer brief intervention-CBI; intervener brief intervention-IBI; enhanced usual care-EUC), and two follow-up conditions (adapted motivational enhancement therapy-AMET; enhanced usual care-EUC) that will take place 3 months post-ED. All individuals who meet criteria for a drug use disorder will additionally receive the "referral to treatment" or "RT" component of SBIRT. Stratified random assignment [by gender and diagnosis of a drug use disorder (yes/no)] will take place at baseline for all ED based and follow-up conditions. All participants will receive written information including substance abuse and other community resources, and HIV prevention materials. Recognizing that brief interventions are important, but not necessarily sufficient, for change in all patients who use drugs, the primary specific aims of the proposed study will determine the independent effectiveness of immediate "on-the-spot" ED-based brief intervention conditions, 3-month followup brief treatment conditions, and combinations of conditions, for decreasing drug use and improving health-related outcomes (including physical and mental health, and HIV risk behavior) at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* patients age 18-60 years presenting to the HMC for medical care (except exclusions as noted below)
* ability to provide informed consent. Additional inclusion criteria for intervention: past 3-month use of illicit drugs or misuse of psychoactive prescription drugs

Exclusion Criteria:

* patients who do not understand English (less than 1% in our prior work) -
* prisoners
* patients classified by medical staff as "Level 1 trauma" (e.g., unconscious, intubated on respirators, in need of immediate lifesaving procedures such as surgery)
* patients deemed unable to provide informed consent as stated above (e.g., intoxication, mental incompetence)
* patients treated in the ED for suicide attempts or sexual assault

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 878 (Actual)
Dates: Start 2011-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
drug use | change over time (3, 6 and 12 months post-baseline)
  Drug use is measured using the NIDA-Modified ASSIST (Alcohol, Smoking and Substance Involvement Screening Test).
drug use - number of days used | change over time (3, 6 and 12 months post-baseline)

SECONDARY OUTCOMES:
HIV risk behaviors | change over time (3, 6 and 12 months post-baseline)
  HIV risk behaviors are measured using the Health Related Behavior Survey (HRBS).
health related outcomes (physical health) | change over time (3, 6 and 12 months post-baseline)
  Physical health is measured using the Short Form Health Survey (SF-12).
health related outcomes (mental health) | change over time (3, 6 and 12 months post-baseline)
  Mental health is measured using the Brief Symptom Inventory (BSI-18).
health related outcomes (mental health) | change over time (3, 6 and 12 months post-baseline)
  Mental health is measured using the Patient Health Questionnaire (PHQ-9).

CONTACTS AND LOCATIONS:
Overall Officials: Frederic C Blow, PhD, Principal Investigator — University of Michigan
Locations (1):
- Hurley Medical Center Emergency Department, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drislane LE, Waller R, Martz ME, Bonar EE, Walton MA, Chermack ST, Blow FC. Therapist and computer-based brief interventions for drug use within a randomized controlled trial: effects on parallel trajectories of alcohol use, cannabis use and anxiety symptoms. Addiction. 2020 Jan;115(1):158-169. doi: 10.1111/add.14781. Epub 2019 Oct 24. PMID 31400240